CLINICAL TRIAL: NCT03225222
Title: MRI in PROstate Cancer Diagnosis With Prior Risk Assessment
Acronym: MR-PROPER
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ivo G. Schoots, Dr., Erasmus Medical Center
Other Study IDs: OZBS92.16132
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; multivariate risk assessment; MRI; biopsy; screening; multicenter
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low-risk PCa: No TRUS-guided biopsy
- Intermediate/high-risk PCa (Control): TRUS-guided biopsy 'only' (current standard practice).
  Interventions: Diagnostic Test: biopsy
- Intermediate/high-risk PCa (Intervention 1): TRUS-guided biopsy 'first'; if indicated followed by MRI and targeted biopsies.
  Interventions: Diagnostic Test: biopsy
- Intermediate/high-risk PCa (Intervention 2): MRI-'first', followed by TRUS-guided and targeted biopsies.
  Interventions: Diagnostic Test: biopsy

INTERVENTIONS:
Diagnostic Test: biopsy — prostate biopsy
  Groups: Intermediate/high-risk PCa (Control); Intermediate/high-risk PCa (Intervention 1); Intermediate/high-risk PCa (Intervention 2)

SUMMARY:
To evaluate the diagnostic performance and cost-effectiveness of the MRI-driven diagnostic pathway of prostate cancer, with upfront individual multivariate risk stratification.

DETAILED DESCRIPTION:
Screening for prostate cancer (PCa) remains one of the most controversial issues in urological practice. Although robust data from the European Randomised study of Screening for Prostate Cancer (ERSPC) suggest a disease specific survival benefit in favor of prostate-specific antigen (PSA)-based PCa screening, the coinciding unfavorable harm-benefit precludes that PCa screening can be adopted as a public health policy. The diagnostic pathway needs to be optimized to reduce unnecessary testing and to avoid diagnosing those cancers that will never harm a patient if not detected through screening. Some men may thus benefit from PCa screening, but with the currently used diagnostics (i.e. the PSA test and systematic TRUS (transrectal ultrasound )-guided prostate biopsy) many more men are harmed by unnecessary testing and the cascade of diagnostic and treatment related events that follow.

Further refinements to screening strategies, focusing on detecting only those PCa that are potentially life threatening (clinically significant) are needed to become acceptable to the general population and health care providers. The investigators propose such a refinement within this protocol, with upfront individual risk prediction and in addition a MRI-driven diagnostic pathway in only those men that are considered to be at intermediate/high-risk of having a potentially life threatening PCa (in general defined as Gleason sum Score (GS) =7).

ELIGIBILITY:
Inclusion criteria:

* men ≥ 50 years,
* no prior prostate biopsies,
* suspected of having prostate cancer based on PSA blood test (≥ 3 ng/ml) and/or DRE( digital rectal examination) and/or family history of prostate cancer,
* fit to undergo all protocol procedures,
* signed informed consent.

Exclusion criteria:

* contra-indications to MRI or TRUS biopsy procedures,
* any medical condition precluding procedures described in the protocol

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men are eligible for the study if there is a clinical suspicion of harbouring prostate cancer without previous prostate biopsies. This essentially includes men with an elevated PSA (≥ 3 ng/ml) and/or a suspicious DRE, or family history of prostate cancer.
Sampling Method: Probability Sample
Enrollment: 2558 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of detected csPCa | 36 months
  Proportion of study population with clinically significant prostate cancer (csPCa), correctly identified by Risk-assessment + MRI-driven pathway

SECONDARY OUTCOMES:
Number of biopsy procedures in relation to detected csPCa. | 36 months
  Number of prostate biopsy procedures in relation to the detection of clinically significant prostate cancer.
Proportion of unnecessary TRUS-guided and targeted biopsies | 36 months
  Proportion of TRUS-guided and targeted biopsies that could have been avoided safely.
CEA Risk stratification-MRI | 36 months
  Diagnostic health care cost-effectiveness analysis (CEA) of Risicowijzer-MRI-driven pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Schoots, Dr, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmusmc, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Still under consideration